CLINICAL TRIAL: NCT05314478
Title: Safe and Effective Headgear Accessory for Exercise-Induced Laryngeal Obstruction Studies (HALOS) - a Device Development Study
Brief Title: Headgear Accessory for Exercise-Induced Laryngeal Obstruction Studies
Acronym: HALOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SP0707
Record Dates: First submitted 2022-03-30; First posted 2022-04-06 (Actual); Results first posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2023-10

CONDITIONS: Exercise-Induced Laryngeal Obstruction
Keywords: Laryngoscopy; Exercise-Induced; Laryngeal Obstruction; Headgear

STUDY DESIGN:
Intervention Model Description: The study is an interventional clinical trial involving a single group of 30 participants undergoing a continuous laryngoscopy during exercise test with the HALOS headgear.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): Participants will be required to attend a single consultation and screening appointment to discuss the investigation procedure, and this will occur at least a week before the Continuous Laryngoscopy during Exercise (CLE) test. Participants will then attend one appointment for the CLE test. There will be no follow up assessments using the headgear.
  Interventions: Device: Continuous laryngoscopy during exercise test using the HALOS headgear

INTERVENTIONS:
Device: Continuous laryngoscopy during exercise test using the HALOS headgear — The participant will undergo the CLE test following standard clinical practice.
  The order of events of the aspects of the investigation related to the headgear will be:
  1. The headgear is prepared for use.
  2. The headgear is fitted onto the participant's head.
  3. The endoscope is inserted into the participant.
  4. The endoscope is fitted onto the headgear.
  5. The CLE test is carried out.
  6. The endoscope is removed from the headgear.
  7. The endoscope is removed from the participant.
  8. The headgear is removed from the participant.
  9. The headgear is cleaned and stored.

SUMMARY:
Exercise-induced laryngeal obstruction (EILO) is a condition in which the larynx, or voice box, narrows during high-intensity exercise, and is often mis-diagnosed. A test called a Continuous Laryngoscopy during Exercise (CLE) test can be performed, where a flexible camera is inserted through the nose and positioned at the back of the throat. While the patient exercises, the camera image can be used to identify the presence of EILO.

During the CLE test it is important that the part of the camera that remains outside the body is held securely in position near the forehead so that a clear and stable image is obtained using a headgear to secure the camera to the patient's head.

There are no headgears available on the market, so we have designed and manufactured one called HALOS (Headgear Accessory for Exercise-Induced Laryngeal Obstruction Studies).

This study is to ensure that HALOS is suitable for use, and to check we have understood and minimised the risks associated with the headgear. The headgear can then be used routinely within the Trust, improving the care that offered to patients.

We will recruit 30 male or female participants who need to undergo a CLE test. The study will be conducted at Broadgreen Hospital, Liverpool, UK. Before the CLE test, participants will attend a screening appointment to discuss the procedure. There will be no follow-up appointments.

During the CLE test, the participants will wear the HALOS headgear while exercising, and the clinician will monitor the image from the camera for signs of EILO. After the test, participants will be asked how tolerable the headgear was, and if they have any concerns about any aspect of it. The clinician will also record how clear and stable the camera image was, how easy it was to use, and any concerns about any aspect of it.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male, female or non-binary, aged 18 years or above.
* Able (in the Investigators opinion) and willing to comply with all study requirements.
* Able to undergo a CLE test as judged by the clinician, and where a clinical need of the test for the delivery of healthcare has been identified.

Exclusion Criteria:

* Pain, sore areas, broken skin at the site of contact with the headgear.
* Devices, e.g. cochlear implants, that impede the use of the headgear.
* Head circumference is less than 50cm or greater than 63cm, reflecting the 3rd centile for females and 97th centile for males, respectively (Bushby, 1992).
* Exclusion criteria for endoscopy procedures:

  * Skull base/facial surgery or fracture within the previous six weeks
  * Major or life threatening epistaxis within the previous six weeks
  * Trauma to nasal cavity secondary to surgery or injury within the previous six weeks
  * Sino-nasal and anterior skull base tumours/surgery
  * Nasopharyngeal stenosis
  * Craniofacial anomalies
  * Hereditary haemorrhagic telangiectasia
  * Severe movement disorders and/or severe agitation
  * Vasovagal history
  * Bleeding risks
* Any other exclusion criteria as identified by the current endoscopy procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tristan Payne, Principal Investigator — Liverpool University Hospitals NHS Foundation Trust
Locations (1):
- Liverpool University Hospitals Nhs Foundation Trust, Liverpool, Merseyside, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants: Participants will be required to attend a single consultation and screening appointment to discuss the investigation procedure, and this will occur at least a week before the Continuous Laryngoscopy during Exercise (CLE) test. Participants will then attend one appointment for the CLE test. There will be no follow up assessments using the headgear.
  Continuous laryngoscopy during exercise test using the HALOS headgear: The participant will undergo the CLE test following standard clinical practice.
  The order of events of the aspects of the investigation related to the headgear will be:
  1. The headgear is prepared for use.
  2. The headgear is fitted onto the participant's head.
  3. The endoscope is inserted into the participant.
  4. The endoscope is fitted onto the headgear.
  5. The CLE test is carried out.
  6. The endoscope is removed from the headgear.
  7. The endoscope is removed from the participant.
  8. The headgear is removed from the participant.
  9. The headgear is cleaned and stored.
Period: Overall Study
Arm/Group | Participants
Started | 30
Completed | 29
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Participants
Number analyzed (Participants) | 29
Age, Continuous [Median (Full Range); unit: years] | 35 [22 to 76]
Sex/Gender, Customized [Count of Participants; unit: Participants] — Sex not collected Population: Sex not collected
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Head circumference [Median (Full Range); unit: centimetres] | 56.5 [52 to 61]
Form of exercise [Count of Participants; unit: Participants]
  Treadmill | 23
  Stationary bike | 6
Scope used [Count of Participants; unit: Participants]
  Ambu aScope 4 RhinoLaryngo endoscope | 26
  XION Video Nasopharyngoscope EV-NC endoscope | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Continuous Laryngoscopy During Exercise Tests
Description: The percentage of participants with continuous laryngoscopy during exercise tests where the endoscopy image was clear and stable enough to allow a diagnosis of exercise-induced laryngeal obstruction to be confirmed or ruled out.
Time Frame: 30 minutes
Measure: Number; unit: percentage of participants
Arm/Group | Participants
Number analyzed (Participants) | 29
percentage of participants | 100

2. Secondary Outcome: Percentage of Participants With Device Usability Rating of 4 or 5
Description: The percentage of participants where the clinician provided a device usability rating of 4 or 5 on the post-test questionnaire. Device usability is scored on a five-point LIKERT scale ranging from 1 (very hard to use) to 5 (very easy to use).
Time Frame: 60 minutes
Measure: Number; unit: percentage of participants
Arm/Group | Participants
Number analyzed (Participants) | 29
percentage of participants | 96.6

3. Secondary Outcome: Device Usability Subjective Feedback
Description: Focussing on any clinician-reported concerns regarding set-up, operation and cleaning.
Time Frame: 60 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Participants
Number analyzed (Participants) | 29
Participants
  Ease of tightening headgear raised as an issue, caused by participant's small head | 1
  Ease of tightening headgear raised as an issue, unknown cause | 2
  Did not comment on usability | 26

4. Secondary Outcome: Percentage of Participants Scoring Device Tolerability as 3 or 4
Description: The percentage of participants where the participant provided a device tolerability rating of 3 or 4 on the post-test questionnaire. Device tolerability is scored on a four-point scale of 1 (highly intolerable), 2 (intolerable), 3 (tolerable) or 4 (highly tolerable).
Time Frame: 60 minutes
Measure: Number; unit: percentage of participants
Arm/Group | Participants
Number analyzed (Participants) | 29
percentage of participants | 100

5. Secondary Outcome: Device Tolerability Subjective Feedback
Description: Focussing on any participant-reported concerns regarding the comfort of the headgear including how hot their head felt, weight of the headgear, how secure the headgear felt and the impact of the headgear on their performance during the investigation.
Time Frame: 60 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Participants
Number analyzed (Participants) | 29
Participants
  Comments related to how heavy the headgear felt: Raised as an issue, but they did did not feel impacted by this when exercising. | 6
  Comments related to how heavy the headgear felt: Raised as an issue, but didn't indicate whether they felt impacted by this when exercising. | 2
  Comments related to how heavy the headgear felt: Commented that this was acceptable. | 11
  Comments related to how heavy the headgear felt: Did not comment on this | 10
  Comments related to how hot their head felt: Raised as an issue, but they did did not feel impacted by this when exercising. | 3
  Comments related to how hot their head felt: Raised as an issue, but didn't indicate whether they felt impacted by this when exercising. | 2
  Comments related to how hot their head felt: Commented that this was acceptable. | 4
  Comments related to how hot their head felt: Did not comment on this | 20
  Comments related to how stable the headgear felt: Raised as an issue, but they did did not feel impacted by this when exercising. | 2
  Comments related to how stable the headgear felt: Raised as an issue, but didn't indicate whether they felt impacted by this when exercising. | 2
  Comments related to how stable the headgear felt: Commented that this was acceptable. | 13
  Comments related to how stable the headgear felt: Did not comment on this | 12

ADVERSE EVENTS:
Time Frame: 30 minutes.
Arm/Group | Participants
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-22): https://cdn.clinicaltrials.gov/large-docs/78/NCT05314478/Prot_SAP_000.pdf